CLINICAL TRIAL: NCT05189483
Title: Albumin-bound Paclitaxel Plus Camrelizumab Therapy in Locally Unresectable or Metastatic Soft Tissue Sarcomas After Failure of First Line Chemotherapy: a Single Institution, Open-label, Phase 2 Trial
Brief Title: Albumin-bound Paclitaxel Plus Camrelizumab for Advanced Soft Tissue Sarcoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Jiaqiang, Doctor, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZZUSC-2
Record Dates: First submitted 2021-12-29; First posted 2022-01-12 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-10

CONDITIONS: Soft Tissue Sarcoma
Keywords: Albumin-bound paclitaxel; Camrelizumab; PD-1; Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Albumin-Bound Paclitaxel; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Albumin-bound paclitaxel plus camrelizumab therapy arm (Experimental): Enrolled patients will receive the following treatment: 300 mg/m2 of nab-paclitaxel (Hengrui Pharmaceutical, Lianyungang, China) and 200 mg of PD-1 inhibitor (camrelizumab; Hengrui Pharmaceutical, Lianyungang, China) via a 30-min intravenous infusion on day 1. The treatment was repeated every three weeks.
  Interventions: Drug: Albumin-Bound Paclitaxel; Drug: Camrelizumab

INTERVENTIONS:
Drug: Albumin-Bound Paclitaxel — Enrolled patients will receive 300 mg/m2 of nab-paclitaxel (Hengrui Pharmaceutical, Lianyungang, China) via a 30-min intravenous infusion on day 1. The treatment was repeated every three weeks until progressive disease occurrence or unacceptable adverse events.
Drug: Camrelizumab — Enrolled patients will receive the following treatment: 200 mg of PD-1 inhibitor (camrelizumab; Hengrui Pharmaceutical, Lianyungang, China) via a 30-min intravenous infusion on day 1. The treatment was repeated every three weeks until progressive disease occurrence or unacceptable adverse events.

SUMMARY:
In this open, single center, one- armed clinical study, enrolled patients will receive the following treatment: 300 mg/m2 of nab-paclitaxel (Hengrui Pharmaceutical, Lianyungang, China) and 200 mg of PD-1 inhibitor (camrelizumab; Hengrui Pharmaceutical, Lianyungang, China) via a 30-min intravenous infusion on day 1. The treatment was repeated every three weeks until progressive disease occurrence or unacceptable adverse events.

The primary end point was progression-free survival at 4 months. Secondary objectives were objective response rate and safety.

DETAILED DESCRIPTION:
There is increasing evidence that combination therapy with nanoparticle albumin-bound paclitaxel (nab-paclitaxel) and programmed cell death protein 1 (PD-1) inhibitor is safe and efficacious in treating many types of malignant tumors. However, clinical data demonstrating the effect of this treatment combination for patients with metastatic soft tissue sarcoma are currently limited.

In this open, single center, one- armed clinical study, enrolled patients will receive the following treatment: 300 mg/m2 of nab-paclitaxel (Hengrui Pharmaceutical, Lianyungang, China) and 200 mg of PD-1 inhibitor (camrelizumab; Hengrui Pharmaceutical, Lianyungang, China) via a 30-min intravenous infusion on day 1. The treatment was repeated every three weeks until progressive disease occurrence or unacceptable adverse events.

The primary end point was progression-free survival at 4 months. Secondary objectives were objective response rate and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 16-70, male and female.
2. ECOG score of physical condition was 0-1. This can be extended to 2 points for amputees.
3. Expected survival ≥3 months.
4. Subjects with distant metastases or locally advanced soft tissue sarcomas determined by the investigator to be unsuitable for surgical treatment (pathologic subtypes include undifferentiated pleomorphic sarcomas, synovial sarcomas, leiomyosarcomas, hemangiosarcomas, clear cell sarcomas, epithelioid sarcomas, fibrosarcomas, and undifferentiated/poorly differentiated liposarcomas).
5. Subjects with metastatic/surgically unresectable soft tissue sarcoma who received prior systemic treatment or who had a sensitive recurrence (a recurrence more than 6 months after the last chemotherapy) after chemotherapy.
6. Measurable lesions in compliance with RECIST1.1 criteria.
7. All acute toxicities resulting from prior antitumor therapy or surgery were alleviated by the first day of the first cycle (C1D1) to level 0-1 (according to NCI-CTCAE 4.03) or to the level specified in the inclusion/exclusion criteria (except for toxicities such as hair loss that the investigator did not consider to pose a safety risk to the subject).
8. Patients must have adequate organ function (without blood transfusion, without growth factor or blood components support within 14 days before enrollment)as determined by: Hemoglobin ≥ 9 g/dL; Absolute neutrophil count (ANC) ≥1.5×109/L; Platelet count ≥ 75×109/L (for patients with advanced hepatocellular carcinoma), Platelet count ≥ 100×109/L (for patients with advanced gastric cancer); serum albumin ≥2.8 g/dL; serum total bilirubin (TBIL)≤1.5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×upper limit of normal(ULN), for subjects with liver metastases, ALT and AST≤5×ULN; Calculated creatinine clearance (CrCl) > 50 mL/min (Cockcroft-Gault formula will be used to calculate CrCl).
9. Urine routine: urine protein <2+; If urine protein ≥2+, 24-hour urine protein quantification must be ≤1g; Thyroid function: Thyroid stimulating hormone (TSH)≤ULN; If FT3(T3) and FT4(T4) levels are abnormal, FT3(T3) and FT4(T4) levels can be selected if they are normal.
10. Female subjects of reproductive age must have performed a serum pregnancy test negative within 7 days prior to medication and be willing to use a medically approved highly effective contraceptive method (e.g., an intrauterine device, birth control pill, or condom) during the study period and for 3 months after the last medication; Male subjects with a female partner of reproductive age were surgically sterilized or agreed to use an effective method of contraception during the study period and for 3 months after the last study administration.
11. With my consent and informed consent, I am willing and able to comply with the planned visit, research treatment, laboratory examination and other experimental procedures.

Exclusion Criteria:

1. Has received the following treatments within the first 4 weeks before C1D1: tumor radiotherapy, surgery, chemotherapy, immunotherapy or molecular targeted therapy; Other investigational drugs; Receive live attenuated vaccine.
2. Prior treatment with PD-1/PD-L1/CTLA-4 antibody.
3. Surgical treatment and/or radiotherapy for soft tissue sarcoma are planned for the study period.
4. Imaging diagnosis showed the presence of tumor lesions in the central nervous system.
5. Prior use of immunosuppressive drugs within 14 days prior to C1D1, excluding nasal spray and inhaled corticosteroids or physiological doses of systemic steroids (i.e., no more than 10mg/ day of prednisolone or other corticosteroid at pharmacophysiological dose).
6. The presence or history of any active autoimmune diseases (including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism); Subjects with vitiligo or asthma that was in complete remission during childhood and did not currently require medical intervention could be included), or a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
7. Severe infection (e.g., antibiotic, antifungal, or antiviral) within 4 weeks prior to C1D1, or unexplained fever >38.5°C during screening/prior to initial administration.
8. Hypertension that cannot be well controlled by antihypertensive medication (systolic blood pressure > 140 mmHg or diastolic blood pressure >90mmHg).
9. Bleeding symptoms with significant clinical significance or clear bleeding tendency occurred within 3 months before C1D1, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occultation blood ++ or above, vasculitis, etc. Or arteriovenous thrombosis events occurring within 6 months prior to C1D1, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.; Or long-term anticoagulant therapy with warfarin or heparin, or long-term antiplatelet therapy (aspirin ≥300mg/ day or clopidogrel ≥75mg/ day).
10. Active heart disease, including myocardial infarction, severe/unstable angina, within 6 months prior to C1D1. Arrhythmias with poorly controlled left ventricular ejection fraction <50% on echocardiography (including QTcF interval >450ms in men and >470ms in women).
11. Has been diagnosed with any other malignancy within the previous 3 years prior to C1D1, except for adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix.
12. Known allergy to the study drug or any excipients thereof; Or severe allergic reactions to other monoclonal antibodies.
13. Human immunodeficiency virus (HIV) infection, active hepatitis B (hbSAG positive and HBV-DNA ≥500IU/ mL), hepatitis C (HCV antibody positive and HCV-RNA higher than the lower limit of detection method).
14. In the investigator's judgment, there are concomitant diseases (e.g., poorly controlled hypertension, severe diabetes, neurological or neurologic diseases, etc.) or any other conditions that seriously endanger the safety of the subjects, may confuse the results of the study, or may interfere with the completion of the study.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Up to approximately 24months
  Progression-free survival is defined as time from enrollment to the first occurrence of progression of disease or death from any cause within 63 days of last response assessment.

SECONDARY OUTCOMES:
Objective response rate | Up to approximately 24months
  Defined as the proportion of patients who achieve partial response or complete response according to RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Bone and Soft Tissue, Henan Cancer Hospital, Zhengzhou, Henan, China